CLINICAL TRIAL: NCT06775197
Title: Sterile Allogeneic Spongioflex® Allograft As Partial Meniscal Replacement After Incomplete Meniscal Loss, an Investigator-initiated Trial
Brief Title: Partial Meniscal Replacement with Spongioflex®
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maria-Josef-Hospital Greven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Spongioflex_EK_5324_01
Record Dates: First submitted 2024-12-23; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Partial Meniscal Loss; Lateral Meniscus Partial Loss; Medial Meniscal Partial Loss; Meniscus Lesion; Meniscal Injuries; Meniscal Tear
Keywords: partial meniscal loss; Allograft; Spongioflex®; IKDC; KOOS; return to sport; Outerbridge score; extrusion; VAS pain score

STUDY DESIGN:
Intervention Model Description: Low interventional trial with 2 arms (operated group in comparison to non-operated group)
Who Masked: Participant
Masking Description: non
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- operated group (partial meniscal replacement) (Active Comparator): Patients, who decide to get operated will be in the experimental group, Spongioflex® will be the investigational product
  Interventions: Procedure: partial meniscal replacement with Spongioflex®
- non-operated patients (No Intervention): Patients who do not decide to be operated at this stage, but want to be closely monitored to eventually join the operated group later.

INTERVENTIONS:
Procedure: partial meniscal replacement with Spongioflex® — for any surgical procedure, the patient receives an antibiotic shot NIMP) just before surgery. The patient will be arthroscopically treated via the arthroscopic portal with implantation of a demineralized bone block (IMP: Spongioflex ®, appropriate size (DIZG gGmbH, Berlin, Germany)) as a partial meniscus substitute. The block will be adapted to the defect size and secured with 2-4 inside-out sutures (Etibond 0, Ethicon, Somerville, NJ). No dosing, the IMP has no systemic effect. The surgery (Intervention) will last between 60-90 minutes. The hospital stay is between 2-3 days after surgery. Follow-up visits: at the end of the hospital stay, after 6 weeks, after 6, 12 and 24 months and after 5 years for the operated group.
  Arms: operated group (partial meniscal replacement)

SUMMARY:
The purpose of this investigator-initiated trial is to evaluate whether the novel graft can prevent/reduce the disadvantages of the previously used replacement materials and shows better results than the group of patients, which were not operated. Since there is currently no alternative made of biological material to this product, this investigator-initiated trial is of great medical and economic importance. The otherwise following arthrosis or knee prosthesis implantation (TKA ) could be prevented or at least postponed. Initial clinical results are promising.

An important and sensitive parameter for assessing the postoperative function of the meniscus is the MRI image. Genovese et al. 2007 were able to show in a categorization/classification which magnetic resonance image can be expected in the case of successful incorporation. Several studies have shown that the known clinical knee scores (Lysholm, IKDC, KOOS, VAS pain) improve significantly after successful ingrowth of the meniscus implant.

DETAILED DESCRIPTION:
The menisci consist of fibrocartilage. They are partially (laterally more than medially) mobile parts of the joint surfaces and compensate for the incongruence of the femur and tibia. They reduce the joint pressure on the tibial plateau and the femoral condyles and help to stabilize the joint. Due to this biomechanical relevance, the partial loss of the meniscus leads to arthritic changes in long term. Suturing the torn meniscus is increasingly becoming the focus of knee surgery. Degenerative torn menisci have a significantly poorer prognosis with regard to healing than traumatically torn menisci (e.g. meniscus damage associated with a cruciate ligament tear).

Indications for partial meniscus replacement are symptomatic, degenerative, and irreparable damage to the medial and lateral meniscus, possibly with early osteoarthritis of the compartments, as well as partial loss of the meniscus in the event of anterior knee instability in young, active patients, in which case simultaneous reconstruction of the anterior cruciate ligament should be performed. A prerequisite for a good clinical result after partial meniscus replacement is a stable knee without malalignment in the coronal plane. Partial meniscus replacement is not suitable in the case of axial deviation and knee instability, patients older than 60 years, advanced chondromalacia and degenerative changes in the affected compartment, an extension deficit of more than 3° compared to the opposite side or a knee flexion of less than 125°. Inflammatory arthritis or synovial inflammation of the knee and a BMI greater than 30 kg/m² are additional exclusion criteria.

Williams et al. 2007 could show, that 5 years after partial removal of the medial or lateral meniscus, despite an excellent functional result, 64% of patients showed medial and 33% lateral cartilage damage on MRI. This study highlights the considerable delay with which the symptoms occur despite already detectable arthritic changes.

Englund et al. were able to show in a study that patients developed osteoarthritis significantly more frequently over a period of 30 months if they had meniscus damage than if they did not. Englund et al. detected tibiofemoral osteoarthritis in 27% of patients 15 years after partial meniscus removal, compared to 10% in a control group that had not undergone surgery.

In the case of incomplete meniscus loss, where the peripheral rim is sufficiently intact, defect filling is the only way to restore the lost substance and function of the meniscus. In the past, an implant made of bovine collagen (Collagen Meniscus Implant (CMI), Stryker) or an artificial meniscus made of polyurethane (Actifit, 2med) was often used. The CMI has been withdrawn from the market by the manufacturer, so that no biological treatment alternative exists.

Schenk et al. were able to show in a recent study for the CMI, consisting of bovine collagen, that, despite a significant improvement in pain and function, the CMI is subject to a progressive shrinkage process over time. The studies mentioned above make it clear that partial replacement of the meniscus is necessary if preservation by meniscus suturing is no longer possible to prevent or postpone arthritic changes.

In the investigator-initiated study on which this application is based, a novel implant made from demineralized allogenic human cancellous bone (Spongioflex®, DIZG gGmbH Berlin) is to be implanted into the meniscus defect of the recipient knee. This transplant has sponge-like properties and therefore facilitates the ingrowth of cells from the surrounding meniscus[16]. The IMP (Spongioflex®) is decalcified and demineralized, it is hard, when dry, but soft when wet. In the knee the conditions are wet, thus it stays soft. It is pliable and can be easily sutured.

The manufacturer (DIZG gGmbH) did a study of cell ingrowth on Spongioflex®. They describe that ingrowth of cells on Spongioflex® was observed after 28 days, and these cells do not ossify.

Scotti et al. summarizes 2013 the knowledge in respect to meniscal repair as follows:

"In the last decade, striving for optimal restoration of meniscal tissue, the orthopedic surgeon's armamentarium has been enriched by the use of biocompatible meniscus scaffold and meniscal allograft transplantation". "However, despite promising short-term results, none of the current strategies have demonstrated regeneration of a functional, long-lasting meniscal tissue and re-establishment of a proper knee homeostasis in the meniscectomised knee". "The rationale for using a cell-free biomaterial to replace part of the meniscus is based on repopulation of the scaffold by the host cells recruited from the synovium and the meniscal remnants, and subsequent tissue ingrowth which renders this approach cell-based after implantation. A mandatory prerequisite is the absence of both knee instability and malalignment".

This section of the paper of Scotti et al. describes exactly the need for a restoration of the meniscus. Furthermore it defines exactly the features of a scaffold:

"A biomaterial used as scaffold for meniscus tissue engineering purposes should present many features. In particular, the ideal meniscal scaffold should be (i) "cell-instructive", promoting cell differentiation and proliferation if cell-seeded, or cell migration if cell-free; (ii) "biomimetic", mimicking architecture, tribology and mechanical features of the native meniscus; (iii) resilient and resistant to withstand mechanical forces acting in the joint while cells produce ECM; (iv) biocompatible, not evoking any foreign-body reaction also with its degradation products; (v) slowly biodegradable allowing to be gradually replaced by biologic tissue; (vi) open, with high porosity, allowing diffusion of nutrients and catabolic substances; and (vii) easy to handle, to be sutured and to be implanted by the surgeon".

Pereira et al. describes that a meniscal implant, either for partial or total replacement should:

"provide the biomechanical properties but also the biological features to replace the loss of native tissue. Moreover, these approaches include possibilities for patient-specific implants of correct size and shape".

Spongioflex® fulfills all these demands described by Dabaghi et al., Scotti et al. and Peirera et al. and it can be adapted in size and shape and thus is at the moment the optimal choice for partial meniscal replacement.

Dickerson et al. describes that "the scaffold must have a high fluid conductance, concomitant with high porosity…. Porosity allows more rapid cell incorporation along the surface and through the thickness of the scaffold, promoting integration with the host tissue." "The scaffold must guide cells to regenerate all four zones of the tissue structure".

This is the case of Spongioflex® it is porose and can guide cells. Scotti et al. proposes 2013 to use CMI for partial meniscal regeneration, but this product is retracted from the market by now, and they describe already the shrinking of the transplant. Knee stability and an aligned knee are a requisite for the study proposed. Dickerson et al. shows that new fibrocartilage tissue is formed on the demineralized end of the allograft. Results of Credille et al. support these findings. It will not be ossified again. Smith et al. describes that "demineralized cancellous bone sponges are Food and Drug Administration-approved and commercially available products that have the potential to provide biologic and biomechanical augments for rotator cuff healing. The sponge can act as a scaffold for cellular attachment and proliferation".

Credille et al. showed in a recent publication that a biphasic interpositional cancellous allograft (BioEnthesis; Sparta BioPharma, Inc., Madison, NJ) can be used for rotator cuff repair. The allograft is "a porous scaffold for endogenous biological factor migration and thus potentially address the lack of enthesis recapitulation at the rotator cuff repair interface… while the demineralized layer supports soft-tissue ingrowth while acting as a "sponge" to hold bone marrow elements at the repair site".

The group around Prof. Moroder from the Charité has used Spongioflex® for glenoid repair. They describe that the transplant does not calcify again. The glenoid is also no bony structure. They got an ethic vote (EA1/039/18) for using the same product in non-bone structures and could show successful restoration of the glenoid.

Sundar et al. describes that the use of demineralized bone matrix increased fibrocartilage when used for augmentation of rotator cuff repair. The used graft (Spongioflex®) provides a scaffold for cell migration of meniscal cells from neighboring parts of the meniscus. The intended study will show that this kind of allograft is suitable for partial meniscal replacement because it allows cell migration and has enough porosity to allow fluid conductance. As described by Wildemann et al. sufficient growth factors are remaining in the demineralized bone matrix (Spongioflex®) to support new fibrocartilage formation. Scotti et al. underlines the importance of growth factors for meniscal regeneration.

In summary from the literature, it can be concluded, that Spongioflex® is an attractive scaffold for partial meniscal repair because it is fully biological, it still has fibrocartilage inductive factors, allows cell migration, fluid conductivity, resists biomechanical forces, does not provoke immunoreactivity, it is adaptable in size and can easily be sutured. Partial meniscus replacement is an established surgical treatment for patients who have undergone partial meniscus removal, to lead to the ingrowth of cells and the regeneration of meniscus-like tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male and female) with:
2. Partial loss of portions of the

   * lateral meniscus and lateral joint line pain OR
   * medial meniscus and medial joint line pain
3. sufficient standing of the peripheral rim, so that the procedure can be performed
4. Age: 18-60 years
5. signed written informed consent to the study and to provide the scientific data in pseudonymized form

Exclusion Criteria:

1. The presence of anterior cruciate ligament insufficiency which is not resolved by reconstruction of the anterior cruciate ligament within 16 weeks after partial meniscal implantation.
2. Axial deviation (>2° varus or valgus)
3. realignment osteotomy not performed within 12 weeks
4. advanced cartilage damage (grade III according to ICRS) and osteoarthrosis in the affected compartment (grade III according to Kellgren and Lawrence [33])
5. Extension deficit of more than 3° compared to the opposite side or a knee flexion of less than 125°
6. inflammatory arthritis or synovitis on the treated knee
7. BMI greater than 30 kg/m²
8. <18 years, >60 years
9. Chronic pain patients
10. only for patients who will be operated:

    1. with increased anaesthesiologic risk, e.g., with known or predicted difficult airway
    2. with increased risk of bleeding
    3. with increased risk of infection
    4. with necrotic, infected, or poorly perfused host sides
    5. history of allergic reactions
    6. acute hypersensitivity reactions to the IMP or any of its excipients
    7. pregnant woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2029-11-05 (Estimated); Study Completion 2031-11-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of the procedure using the KOOS Score | at 6 weeks, 6 and 12 months (operated patients) and at 2 years and 5 years
  Improvement of KOOS 2 and 5 years after surgery compared to scores of the non-operated group and compared to pre-surgery scores
To evaluate efficacy of the procedure using the IKDC | at 6 weeks, 6 and 12 months (operated patients) and at 2 years and 5 years
  Improvement of IKDC 2 and 5 years after surgery compared to scores of the non-operated group and compared to pre-surgery scores
To evaluate efficacy of the procedure using the VAS pain Score | at 6 weeks, 6 and 12 months (operated patients) and at 2 years and 5 years
  Improvement of VAS pain Score 2 and 5 years after surgery compared to scores of the non-operated group and compared to pre-surgery scores

SECONDARY OUTCOMES:
Safety of the patient using the number of adverse events an serious adverse events | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  Type, frequency and severity of treatment-related AEs and SAEs
Efficacy of the procedure to prevent/prolonge progression to TKA | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  How many patients show a progression of osteoarthrosis up to TKA?
MRI evaluation using outerbridge graduation | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  Outerbridge graduation at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years, comparison between the operated and the non-operated group
MRI evaluation for size of meniscus | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  size of meniscus, at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years, comparison between the operated and the non-operated group
MRI evaluation for number of patients with extrusion | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  number of patients with extrusion at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years, comparison between the operated and the non-operated group
MRI evaluation evaluating the size of extrusion | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  Size of extrusion at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years, comparison between the operated and the non-operated group
Patient satisfaction using a questionnaire | at 6 weeks, 6 and 12 months (for operated patients) and at 2 and 5 years
  Very pleased, pleased, not pleased, very unsatisfied in the operated group after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Kösters, PD, Dr. med, Principal Investigator — Maria-Josef-Hospital Greven GmbH
Locations (1):
- Maria-Josef-Hospital Greven GmbH, Greven, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of rheumatoid arthritis. Ann Rheum Dis. 1957 Dec;16(4):485-93. doi: 10.1136/ard.16.4.485. No abstract available. PMID 13498603
- [Background] Genovese E, Angeretti MG, Ronga M, Leonardi A, Novario R, Callegari L, Fugazzola C. Follow-up of collagen meniscus implants by MRI. Radiol Med. 2007 Oct;112(7):1036-48. doi: 10.1007/s11547-007-0204-y. Epub 2007 Oct 21. English, Italian. PMID 17952676
- [Background] Behrendt S. MRI follow up of bilateral partial meniscal substitution with a demineralized bone block. A case report. Radiol Case Rep. 2022 Oct 27;18(1):21-26. doi: 10.1016/j.radcr.2022.09.091. eCollection 2023 Jan. PMID 36324835
- [Background] Bulgheroni P, Murena L, Ratti C, Bulgheroni E, Ronga M, Cherubino P. Follow-up of collagen meniscus implant patients: clinical, radiological, and magnetic resonance imaging results at 5 years. Knee. 2010 Jun;17(3):224-9. doi: 10.1016/j.knee.2009.08.011. Epub 2009 Oct 2. PMID 19800801
- [Background] Stone KR, Rodkey WG, Webber R, McKinney L, Steadman JR. Meniscal regeneration with copolymeric collagen scaffolds. In vitro and in vivo studies evaluated clinically, histologically, and biochemically. Am J Sports Med. 1992 Mar-Apr;20(2):104-11. doi: 10.1177/036354659202000202. PMID 1558234
- [Background] Zaffagnini S, Marcheggiani Muccioli GM, Lopomo N, Bruni D, Giordano G, Ravazzolo G, Molinari M, Marcacci M. Prospective long-term outcomes of the medial collagen meniscus implant versus partial medial meniscectomy: a minimum 10-year follow-up study. Am J Sports Med. 2011 May;39(5):977-85. doi: 10.1177/0363546510391179. Epub 2011 Feb 4. PMID 21297005
- [Background] Monllau JC, Gelber PE, Abat F, Pelfort X, Abad R, Hinarejos P, Tey M. Outcome after partial medial meniscus substitution with the collagen meniscal implant at a minimum of 10 years' follow-up. Arthroscopy. 2011 Jul;27(7):933-43. doi: 10.1016/j.arthro.2011.02.018. Epub 2011 May 31. PMID 21621373
- [Background] Wildemann B, Kadow-Romacker A, Pruss A, Haas NP, Schmidmaier G. Quantification of growth factors in allogenic bone grafts extracted with three different methods. Cell Tissue Bank. 2007;8(2):107-14. doi: 10.1007/s10561-006-9021-0. Epub 2006 Oct 25. PMID 17063261
- [Background] Wildemann B, Kadow-Romacker A, Haas NP, Schmidmaier G. Quantification of various growth factors in different demineralized bone matrix preparations. J Biomed Mater Res A. 2007 May;81(2):437-42. doi: 10.1002/jbm.a.31085. PMID 17117475
- [Background] Hui PW, Leung PC, Sher A. Fluid conductance of cancellous bone graft as a predictor for graft-host interface healing. J Biomech. 1996 Jan;29(1):123-32. doi: 10.1016/0021-9290(95)00010-0. PMID 8839025
- [Background] Sundar S, Pendegrass CJ, Blunn GW. Tendon bone healing can be enhanced by demineralized bone matrix: a functional and histological study. J Biomed Mater Res B Appl Biomater. 2009 Jan;88(1):115-22. doi: 10.1002/jbm.b.31157. PMID 18683228
- [Background] Smith MJ, Pfeiffer FM, Cook CR, Kuroki K, Cook JL. Rotator cuff healing using demineralized cancellous bone matrix sponge interposition compared to standard repair in a preclinical canine model. J Orthop Res. 2018 Mar;36(3):906-912. doi: 10.1002/jor.23680. Epub 2017 Aug 29. PMID 28792082
- [Background] Credille KT, Wang ZRC, Horner NS, Regan DP, Gadomski BC, Easley JT, Garrigues GE, Yanke AB. Biphasic Interpositional Allograft for Rotator Cuff Repair Augmentation Is Safe in an Ovine Model. Arthroscopy. 2023 Sep;39(9):1983-1997. doi: 10.1016/j.arthro.2023.03.018. Epub 2023 Mar 29. PMID 37001743
- [Background] Dickerson DA, Misk TN, Van Sickle DC, Breur GJ, Nauman EA. In vitro and in vivo evaluation of orthopedic interface repair using a tissue scaffold with a continuous hard tissue-soft tissue transition. J Orthop Surg Res. 2013 Jun 19;8:18. doi: 10.1186/1749-799X-8-18. PMID 23782505
- [Background] Pereira H, Fatih Cengiz I, Gomes S, Espregueira-Mendes J, Ripoll PL, Monllau JC, Reis RL, Oliveira JM. Meniscal allograft transplants and new scaffolding techniques. EFORT Open Rev. 2019 Jun 3;4(6):279-295. doi: 10.1302/2058-5241.4.180103. eCollection 2019 Jun. PMID 31210969
- [Background] Scotti C, Hirschmann MT, Antinolfi P, Martin I, Peretti GM. Meniscus repair and regeneration: review on current methods and research potential. Eur Cell Mater. 2013 Sep 23;26:150-70. doi: 10.22203/ecm.v026a11. PMID 24057873
- [Background] Dabaghi M, Eras V, Kaltenhaeuser D, Ahmed N, Wildemann B. Allografts for partial meniscus repair: an in vitro and ex vivo meniscus culture study. Front Bioeng Biotechnol. 2023 Oct 12;11:1268176. doi: 10.3389/fbioe.2023.1268176. eCollection 2023. PMID 37901839
- [Background] Schenk L, Bethge L, Hirschmann A, Berbig R, Luthi U, Arnold MP, Hirschmann MT. Ongoing MRI remodeling 3-7 years after collagen meniscus implantation in stable knees. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1099-1104. doi: 10.1007/s00167-019-05714-w. Epub 2019 Sep 18. PMID 31535191
- [Background] Rodkey WG, DeHaven KE, Montgomery WH 3rd, Baker CL Jr, Beck CL Jr, Hormel SE, Steadman JR, Cole BJ, Briggs KK. Comparison of the collagen meniscus implant with partial meniscectomy. A prospective randomized trial. J Bone Joint Surg Am. 2008 Jul;90(7):1413-26. doi: 10.2106/JBJS.G.00656. PMID 18594088
- [Background] Englund M, Guermazi A, Roemer FW, Aliabadi P, Yang M, Lewis CE, Torner J, Nevitt MC, Sack B, Felson DT. Meniscal tear in knees without surgery and the development of radiographic osteoarthritis among middle-aged and elderly persons: The Multicenter Osteoarthritis Study. Arthritis Rheum. 2009 Mar;60(3):831-9. doi: 10.1002/art.24383. PMID 19248082
- [Background] Williams RJ 3rd, Warner KK, Petrigliano FA, Potter HG, Hatch J, Cordasco FA. MRI evaluation of isolated arthroscopic partial meniscectomy patients at a minimum five-year follow-up. HSS J. 2007 Feb;3(1):35-43. doi: 10.1007/s11420-006-9031-2. PMID 18751768
- [Background] Cannon WD Jr, Vittori JM. The incidence of healing in arthroscopic meniscal repairs in anterior cruciate ligament-reconstructed knees versus stable knees. Am J Sports Med. 1992 Mar-Apr;20(2):176-81. doi: 10.1177/036354659202000214. PMID 1558246
- [Background] Barrett GR, Field MH, Treacy SH, Ruff CG. Clinical results of meniscus repair in patients 40 years and older. Arthroscopy. 1998 Nov-Dec;14(8):824-9. doi: 10.1016/s0749-8063(98)70018-0. PMID 9848593
- [Background] Papalia R, Franceschi F, Diaz Balzani L, D'Adamio S, Maffulli N, Denaro V. Scaffolds for partial meniscal replacement: an updated systematic review. Br Med Bull. 2013;107:19-40. doi: 10.1093/bmb/ldt007. Epub 2013 Mar 1. PMID 23457205
- [Background] Hoser C, Fink C, Brown C, Reichkendler M, Hackl W, Bartlett J. Long-term results of arthroscopic partial lateral meniscectomy in knees without associated damage. J Bone Joint Surg Br. 2001 May;83(4):513-6. doi: 10.1302/0301-620x.83b4.11364. PMID 11380121
- [Background] Andersson-Molina H, Karlsson H, Rockborn P. Arthroscopic partial and total meniscectomy: A long-term follow-up study with matched controls. Arthroscopy. 2002 Feb;18(2):183-9. doi: 10.1053/jars.2002.30435. PMID 11830813
- [Background] FAIRBANK TJ. Knee joint changes after meniscectomy. J Bone Joint Surg Br. 1948 Nov;30B(4):664-70. No abstract available. PMID 18894618
- [Background] Petty CA, Lubowitz JH. Does arthroscopic partial meniscectomy result in knee osteoarthritis? A systematic review with a minimum of 8 years' follow-up. Arthroscopy. 2011 Mar;27(3):419-24. doi: 10.1016/j.arthro.2010.08.016. Epub 2010 Dec 3. PMID 21126847
- [Background] Ahmed AM, Burke DL. In-vitro measurement of static pressure distribution in synovial joints--Part I: Tibial surface of the knee. J Biomech Eng. 1983 Aug;105(3):216-25. doi: 10.1115/1.3138409. PMID 6688842
- [Background] OUTERBRIDGE RE. The etiology of chondromalacia patellae. J Bone Joint Surg Br. 1961 Nov;43-B:752-7. doi: 10.1302/0301-620X.43B4.752. No abstract available. PMID 14038135